CLINICAL TRIAL: NCT02017184
Title: Non-invasive Sensor for Core Temperature Measurement
Acronym: Drager
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Barliz Adato, head investigator of Heller institute of physiology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-13-0737-BA-CTIL; IDF-1233-2013 (Other: IDF)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Body Temperature Regulation
Keywords: Body Temperature Regulation Sensor Noninvasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Research arm (Experimental): This trial contains one group which will undergo the described protocol while connected to both sensors: a rectal thermistor and a non invasive thermistor.
  Interventions: Biological: Noninvasive core temperature thermistor

INTERVENTIONS:
Biological: Noninvasive core temperature thermistor

SUMMARY:
Soldiers are required to perform and maintain alertness in difficult environmental conditions. The sensor examined in this trail may indicate body core temperature elevation during exertion. 12 male volunteers will arrive to our lab and perform a protocol of sitting and walking in thermoneutral and hot environments with two core temperature sensors. The results obtained from them will be compared.

DETAILED DESCRIPTION:
During the protocol the volunteers will sit in thermoneutral condition for 30 minutes, than they will sit in hot chamber (40 celsius and 40% relative humidity). Afterwards, the participants will walk on a treadmill in 5 km/hr and 4% incline for one hour. The participants will be connected to rectal thermistor which is considered the "gold standard" and to the new noninvasive sensor which is attached to the skin surface.

ELIGIBILITY:
Inclusion Criteria:

* age 18-25 - healthy
* after medical checkup
* after signing concent form
* with no heat stroke medical history

Exclusion Criteria:

* heat stroke medical history
* heart disease
* diabetes
* obesity

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Rectal temperature | 1 year
  The participants will undergo the described protocol and their rectal temperature will be measured by rectal thermistor and the new noninvasive thermistor and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Epstein, PhD, Study Director — Heller institute, Sheba medical center
Locations (1):
- Sheba medical center, Tel-Hashomer, Ramat- Gan, Israel